CLINICAL TRIAL: NCT06983769
Title: Cognition Recovery in Sleep Apnea Patients With Cardiovascular Risk by Evaluating Nasal CPAP Versus Dental Oral Appliance
Brief Title: CPAP vs MAD for OSA in Patients With Cognitive Impairment. A Randomized Clinical Trial
Acronym: CRESCENDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); Ng Teng Fong General Hospital (Other); Alexandra Hospital (Other); National University Heart Centre, Singapore (Other); The University of Sydney, Sydney, Australia (Unknown)
Responsible Party: Principal Investigator, Cardiac, Professor of Medicine, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECOS. 2024-3614
Record Dates: First submitted 2025-04-22; First posted 2025-05-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea (OSA); Mild Cognitive Impairment
Keywords: Sleep, Cognition, Mandibular advancement device, CPAP, Clinical trial,
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Masking Description: Investigators responsible for conducting the MoCA, quality of life questionnaires, and reading the MRI brain will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP arm (Active Comparator): CPAP stands for Continuous Positive Airway Pressure. It is the standard treatment for obstructive sleep apnea (OSA). A CPAP machine delivers a constant stream of air through a mask worn over the nose or nose and mouth during sleep. This air pressure keeps the airway open, preventing pauses in breathing caused by airway collapse.
  CPAP is highly effective, especially for moderate to severe OSA, but some patients may find it uncomfortable or difficult to tolerate.
  Interventions: Device: CPAP
- MAD (Experimental): MAD stands for Mandibular Advancement Device. It is a custom-fitted oral appliance used primarily to treat obstructive sleep apnea (OSA) and snoring. The device works by gently advancing the lower jaw (mandible) forward, which helps keep the airway open during sleep by preventing the tongue and soft tissues from collapsing and blocking the airway.
  MADs are a non-invasive alternative to CPAP therapy and are especially suitable for patients with mild to moderate OSA or those who are intolerant to CPAP.
  Interventions: Device: MAD

INTERVENTIONS:
Device: MAD — Mandibular Advancement Device. It is a custom-fitted oral appliance used primarily to treat obstructive sleep apnea (OSA) and snoring. The device works by gently advancing the lower jaw (mandible) forward, which helps keep the airway open during sleep by preventing the tongue and soft tissues from collapsing and blocking the airway.
  MADs are a non-invasive alternative to CPAP therapy and are especially suitable for patients with mild to moderate OSA or those who are intolerant to CPAP
  Arms: MAD
Device: CPAP — CPAP stands for Continuous Positive Airway Pressure. It is the standard treatment for obstructive sleep apnea (OSA). A CPAP machine delivers a constant stream of air through a mask worn over the nose or nose and mouth during sleep. This air pressure keeps the airway open, preventing pauses in breathing caused by airway collapse.
  CPAP is highly effective, especially for moderate to severe OSA, but some patients may find it uncomfortable or difficult to tolerate.
  Arms: CPAP arm

SUMMARY:
Obstructive sleep apnea (OSA) is a prevalent condition that significantly impacts the sleep health and overall well-being of millions of adults worldwide. It is characterized by breathing difficulties during sleep caused by an obstructed upper airway, leading to fragmented sleep, oxygen deprivation, and increased sympathetic activity. OSA and its associated health problems contribute to an annual economic burden exceeding $150 billion in the United States. Studies have shown that individuals with OSA are 26% more likely to develop cognitive impairment compared to those without the condition. However, despite the effectiveness of continuous positive airway pressure (CPAP) therapy, many patients struggle with acceptance and adherence to this treatment. As an alternative, mandibular advancement devices (MADs) have gained acceptance among OSA patients by improving upper airway anatomy through repositioning of the jaw and tongue, thus reducing collapsibility. This non-invasive approach shows promise, particularly in addressing the unique craniofacial features commonly found in East Asian OSA patients.

To further investigate the efficacy of MAD versus CPAP therapy, a multi-center, randomized clinical trial is proposed. The trial aims to evaluate cognitive function using established assessment tools and explore the relationship between different Asian ethnicities and changes in cognitive function, ambulatory blood pressure, and cerebral oxygen saturation. Additionally, brain MRI will be utilized to examine whether baseline brain structure and function can predict treatment response in OSA patients. Participants diagnosed with moderate-to-severe OSA will be randomly assigned to either the MAD or CPAP group in a 1:1 ratio. Baseline assessments, along with six-month and one-year follow-ups, will be conducted to assess the impact of the interventions. This trial seeks to provide valuable insights into the effectiveness of MAD versus CPAP therapy in Asian populations, specifically focusing on their effects on cognitive function and other relevant outcomes in individuals with OSA.

DETAILED DESCRIPTION:
Aim #1: The primary objective is to compare the effectiveness of MAD and CPAP in improving cognitive function in participants with OSA and cardiovascular risk. The key endpoints of the trial will include cognitive function using the Montreal Cognitive Assessment (MoCA). Participants diagnosed with moderate-to-severe OSA, mild cognitive impairment, and cardiovascular risk will be randomly assigned to either the MAD or CPAP group (1:1). Baseline assessments, along with six- and twelve-month follow-ups, will include the administration of the MoCA. The analysis of covariance (ANCOVA) will be used to compare the between-group differences in the changes observed in various measures of cognitive function. We hypothesize that MAD is non-inferior to CPAP in improving cognitive function.

Aim #2: The second objective is to examine whether brain structural and functional integrity at baseline can predict cognitive recovery after OSA treatment. Besides traditional brain macrostructural measures (grey matter volume, cortical thickness, and white matter hyperintensity), we hypothesize that brain microstructural and functional measures at baseline capturing individual differences in cerebral blood flow (via perfusion), cerebrovascular damage (via diffusion-derived freewater in both grey matter and white matter), functional network in higher-order cognitive networks (via task-free fMRI), and blood-brain barrier integrity (diffusion-prepared perfusion) will predict post-treatment cognition in OSA patients (see Preliminary work).

Aim #3: To understand the relative contribution of the complex disease pathophysiology of OSA and its treatment in cognitive function. We aim to understand the relative contribution of the complex disease pathophysiology of OSA and its treatment in cognitive function. We will explore the relationship between improvement in MoCA score from baseline to 12 months follow-up and the following parameters (1) OSA pathophysiology: Epworth Sleepiness Scale, apnea-hypopnea index, oxygen desaturation index, time with SpO2<90% (T90), arousal index. (2) OSA treatment with CPAP/MAD: CPAP/MAD device adherence

ELIGIBILITY:
Inclusion Criteria:

Age of at least 45 Chinese, Malay, Indian Referred to the sleep clinics of the CRESCENDO participating centers for suspected OSA, underwent a clinically indicated level 1 polysomnography, and diagnosed to have moderate-to-severe OSA (AHI ≥ 15 events/hour) Mild cognitive impairment: MoCA score <27 (for those with >10 years of education) and <26 (for those with ≤10 years of education) Agree to follow the study protocol

Exclusion Criteria:

Known OSA and already on regular treatment Severe cognitive impairment (MoCA <10) Severe hypoxemia on polysomnography ODI >60 or min SpO2 <60% Known schizophrenia, bipolar disorder, severe depression, drug abuse or alcohol abuse Contraindications to MAD: less than six teeth in each arch; inability to advance the mandible and open the jaw widely. Pre-existing temporomandibular joint problems, severe bruxism, and advanced periodontal disease Limited life expectancy (< one year) Cardiac or cerebrovascular events leading to hospitalization in the past three months Complex cardiovascular diseases: cyanotic congenital heart disease, moderate to severe pulmonary hypertension On regular medications that could affect the neurocognitive function and/or alertness

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline, 6 months (primary endpoint), and 12 months
  A score for cognitive function

SECONDARY OUTCOMES:
Ambulatory Blood Pressure | Baseline, 6 months and 12 months
  Blood Pressure
Epworth Sleepiness Scale | Baseline, 6 months and 12 months
  Measure of daytime sleepiness
Sleep Apnea Quality of Life Index (SAQLI) | Baseline, 6 months and 12 months
  Sleep-related quality of life
EQ-5D-5L | Baseline, 6 months and 12 months
  Generic health-related quality-of-life measure across five domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), enhanced with four bolt-on items relevant to sleep and cardiovascular health, and a visual analogue scale (VAS) for self-rated health.
Residual AHI | Baseline, 6 months and 12 months
  Residual AHI is a measure of treatment effectiveness. Trial participants will undergo overnight sleep studies at baseline (pre-treatment), 6-month, and 12-month follow-up.
Device adherence | 6 months and 12 months
  Device adherence will be monitored based on the adherence sensors of the MAD and CPAP
Biomarkers | Baseline, 6 months, 12 months
  NT-pro-BNP, high-sensitivity C-reactive protein, and high-sensitivity troponin, angiopoietin-2, Tie-2, Eselectin, vascular endothelial growth factor [VEGF-A]), and Soluble receptor of advanced glycation endproducts [sRAGE]

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hang Ronald Lee, MBBS, MD, Principal Investigator — National University Heart Centre, Singapore
Locations (1):
- National University Hospital, Kent Ridge, Please Select, Singapore

IPD SHARING:
Plan to Share IPD: No